CLINICAL TRIAL: NCT00649766
Title: Tailored Messages to Increase Eye Examination Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Nancy Ellish, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01EY015899 (NIH); R01EY015899 (NIH)
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Eye Disease; Eye Care
Keywords: tailored health messages; glaucoma; diabetic retinopathy; dilated fundus exams; health behavior
MeSH Terms: conditions — Eye Diseases; Glaucoma; Diabetic Retinopathy; Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): tailored print messages to encourage eye examination behavior
  Interventions: Behavioral: tailored newsletter
- 2 (Active Comparator): targeted print messages to encourage eye examination behavior
  Interventions: Behavioral: targeted newsletter

INTERVENTIONS:
Behavioral: tailored newsletter — Tailored newsletter that addresses each person's stage of change, barriers to getting eye exams, and knowledge of eye exams and eye disease
  Arms: 1
Behavioral: targeted newsletter — Targeted newsletter that contains messages about barriers to getting eye exams and presents facts about glaucoma and African-Americans.
  Arms: 2

SUMMARY:
The purpose of this project is to test two different types of health messages, one that is developed for a specific group (targeted) and the other that is more personalized to individuals (tailored), to see which is better at changing how often people have their eyes examined. We hypothesize that people who get the tailored messages will be more likely to get a dilated eye exam than people who receive the targeted messages.

DETAILED DESCRIPTION:
Studies have shown that people are not getting their eyes examined on a regular basis, even though dilated eye exams can detect eye diseases like glaucoma and diabetic retinopathy early, before significant vision loss has developed. Early detection can lead to earlier treatment, which can save sight by preventing or slowing the progression of these eye diseases. In this project we designed, implemented, and are now evaluating tailored and targeted print health messages to increase eye examination behavior in an African-American population 65 years of age and older, a group at increased risk of glaucoma and diabetes.

ELIGIBILITY:
Inclusion Criteria:

* African-American
* 65 years of age or older
* no dilated fundus exam in past 2 years

Exclusion Criteria:

* appointment for dilated fundus exam scheduled
* no access to phone

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 330 (Actual)
Dates: Start 2006-06; Primary Completion 2008-05 (Estimated); Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
doctor-confirmed dilated eye examination | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J. Ellish, DrPH, MSPH, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Result] Ellish NJ, Royak-Schaler R, Passmore SR, Higginbotham EJ. Knowledge, attitudes, and beliefs about dilated eye examinations among African-Americans. Invest Ophthalmol Vis Sci. 2007 May;48(5):1989-94. doi: 10.1167/iovs.06-0934. PMID 17460251
- [Derived] Ellish NJ, Royak-Schaler R, Higginbotham EJ. Tailored and targeted interventions to encourage dilated fundus examinations in older African Americans. Arch Ophthalmol. 2011 Dec;129(12):1592-8. doi: 10.1001/archophthalmol.2011.190. PMID 22159679